CLINICAL TRIAL: NCT06065969
Title: Photobiomodulation Dosimetry Based on Anthropometric and Hemodynamic Variables in Patients With Orofacial Pain
Brief Title: Photobiomodulation Dosimetry s in Patients With Orofacial Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, Principal Researcher, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBM
Record Dates: First submitted 2023-09-12; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Orofacial Pain; Tension-Type Headache
Keywords: orofacial pain; Tension-Type Headache; photobiomodulation
MeSH Terms: conditions — Facial Pain; Tension-Type Headache | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Local photobiomodulation (Active Comparator): Delivering an energy of 6J per point (60 seconds) at 2 points in the masseter muscle region, 1 point in the temporal muscle, and 1 point in the trapezius muscle in the cervical region. The total application will take 4 minutes per session
  Interventions: Radiation: Photobiomodulation
- Vascular photobiomodulation (Experimental): 660 nm and 100 mW, directing the light beam towards the radial artery region, for 10 minutes per session. The participant will be seated in a comfortable chair with side support for resting their arms during the application
  Interventions: Radiation: Photobiomodulation
- sham local photobiomodulation (Sham Comparator): The same procedures described for local photobiomodulation will be followed; however, the equipment will emit only the sound signal, exactly like the equipment used in local photobiomodulation group, without emitting laser light.
  Interventions: Radiation: Photobiomodulation
- Sham Vascular photobiomodulation (Sham Comparator): The same procedures described for vascular photobiomodulation will be followed; however, the equipment will emit only the sound signal, exactly like the equipment used in vascular photobiomodulation group, without emitting laser light
  Interventions: Radiation: Photobiomodulation

INTERVENTIONS:
Radiation: Photobiomodulation — 660 nm and 100 mW, directing the light beam towards the radial artery region, for 10 minutes per session.

SUMMARY:
This project aims to validate a dosimetry model for photobiomodulation treatment in patients with orofacial pain and tension-type headache symptoms. The study will involve 240 participants divided into four age groups. Different treatment approaches will be applied, including local photobiomodulation and systemic laser therapy. Various physiological measurements will be taken before, during, and after the treatments, including skin type, weight, height, blood pressure, and heart rate. Additionally, data from questionnaires on pain and headache symptoms will be analyzed. Monte Carlo simulation will be employed to validate the model based on these measurements and light transmission. The research addresses the need for effective pain management strategies in cases where medication-based treatments may have unwanted side effects.

ELIGIBILITY:
Inclusion Criteria Individuals of both sexes, between 7 and 65 years of age Exclusion Criteria

Participants with the following characteristics will be excluded:

Pregnant individuals Individuals with arrhythmia Individuals with Thrombocytopenia Individuals with Sickle Cell Anemia Individuals with a pacemaker Individuals with alterations in coagulation factors

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Headache and orofacial pain | two weeks
  Headache and orofacial pain assessed using the Visual Analog Scale from zero to 10.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuler SSV, Campos MCV, Lacerda AJ, Mazzoni AC, Silva T, Silva FCD, Martins MD, Fernandes KPS, Fonseca ES, Mesquita-Ferrari RA, Horliana ACRT, Bussadori SK, Motta LJ. Dosimetry model for photobiomodulation based on anthropometric and hemodynamic variables in patients with orofacial pain post-Covid-19: Study protocol for randomized clinical trial. PLoS One. 2024 Oct 15;19(10):e0309073. doi: 10.1371/journal.pone.0309073. eCollection 2024. PMID 39405292